CLINICAL TRIAL: NCT06065111
Title: Study of Osteogenesis Imperfecta Tendon and Ligament: Retrospective and Prospective Assessment.
Brief Title: Study of Osteogenesis Imperfecta Tendon
Acronym: SOIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Hopital Lariboisière (Other); University Hospital, Lille (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: SOIT
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study tendon damage in osteogenesis imperfecta patients: The study will be conducted in three centers: Brussels (30 patients, clinique Saint-Luc, Lille (30 patients) and Paris (50 patients). Patients will be recruited regardless of their form of osteogenesis imperfecta.
  Interventions: Other: study tendon damage in osteogenesis imperfecta patients

INTERVENTIONS:
Other: study tendon damage in osteogenesis imperfecta patients — * To identify and characterize alterations of tendons and ligaments in patients with osteogenesis imperfecta (OI) and to improve clinical management of the disease.
  * To analyze interactions of different parameters, such as laxity or administration of bisphosphonates, on the evolution of the disease.

SUMMARY:
Osteogenesis imperfecta (OI) is a rare genetic disease due to a mutation in one of the genes encoding either type I collagen or a protein involved in its synthesis. This leads to bone fragility with fractures and deformities. However, other tissues rich in type I collagen can also be affected, such as teeth or vessel walls.

In the literature, several case reports describe tendon ruptures in OI patients, but no original study has really addressed this issue, which is likely to impact the quality of life through a reduction in mobility and pain.

Recent work carried out by the investigators shows an alteration of the osteotendinous unit in the osteogenesis imperfecta mouse (oim), a validated model of the most severe form of OI. Consequently, the project aims to study the damage of tendon and ligament in patients suffering from osteogenesis imperfecta.

DETAILED DESCRIPTION:
This project aims to study the damage of tendon and ligament in a cohort of patients suffering from osteogenesis imperfecta. The data collected will be put into perspective with those of our first experimental work on mice. They will also make it possible to complete the specific care of these patients. Indeed, during the anamnesis, particular attention will be paid to the description of tendon-ligament pain in order to propose the most effective treatment for this kind of disorder, mainly in physiotherapy. Prevention work will surely be necessary with patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* to have an osteogenesis imperfecta

Exclusion Criteria:

* none, since we want to study different types of osteogenesis imperfecta and consider the effect of age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with osteogenesis imperfecta
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Tendon stiffness | Throughout the entire study, approximately during 22 months
  Triceps suralis tendon, from zero to infinity, expressed in Newton/mm², a high value indicates a high stiffness

SECONDARY OUTCOMES:
Grip strength test | Throughout the entire study, approximately during 22 months
  Dynamometer
Kinesiophobia | Throughout the entire study, approximately during 22 months
  Tampa questionnaire
Mobility : walking test | Throughout the entire study, approximately during 22 months
  Timed-up and go (if walking is possible for the patient)
Quality of life for children | Throughout the entire study, approximately during 22 months
  Pediatric Quality of Life Inventory
Quality of life for adults | Throughout the entire study, approximately during 22 months
  Medical Outcomes Study 36-item Short-Form Health Survey
Pain localization and intensity for children | Throughout the entire study, approximately during 22 months
  face scale
Pain localization and intensity for adults | Throughout the entire study, approximately during 22 months
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Louis Docquier, MD, Principal Investigator — Cliniques Univresitaires Saint-Luc
Locations (1):
- Pole de Morphologie, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No